CLINICAL TRIAL: NCT04380181
Title: Does the Choice of Perioperative Inotropes Has Influence on the Morbidity and Mortality of Infants Operated for Complex Heart Defects?
Brief Title: Influence of Inotropic Choice on Morbidity and Mortality in Complex Pediatric Heart Surgery
Acronym: CHUBpedCSino
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Collaborators: Queen Fabiola Children's University Hospital (Other)
Responsible Party: Principal Investigator, Denis SCHMARTZ, Head, Anesthesiology, Brugmann University Hospital
Other Study IDs: CHUB-ped_CS_inotropes
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Pediatric Cardiac Surgery
Keywords: pediatric cardiopulmonary bypass; milrinone; dobutamine; epinephrine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dobutamine: Weaning from cardiopulmonary bypass using dobutamine as inotrope.
  Interventions: Drug: dobu
- Milrinone-epinephrine: Weaning from cardiopulmonary bypass using milrinone and epinephrine as inotropes.

INTERVENTIONS:
Drug: dobu — Use of dobutamine versus milrinone and epinephrine for separation from cardiopulmonary bypass
  Other Names: milrinone-epinephrine
  Groups: Dobutamine

SUMMARY:
Our study is based on the observation that management of the cardiopulmonary by-pass withdrawal in pediatric heart surgery is quite variable between medical teams.

Indeed, in our center (HUDERF), the most common inotropic plan is dobutamine only or combination of milrinone and adrenalin but their uses seem to be very anesthesiologist dependent.

Despite the lack of sufficient evidence, the choice is probably multi-factorial, based mainly on the inotrope pharmacology, the patient physiopathology and the anesthesiologist preference.

The aim of this study is to determine if one of these inotropic strategy (dobutamine VS milrinone + adrenaline) is better compared to the other in terms of morbi-mortality.

In order to do that, the investigators will realize a retrospective study based on files from January 2008 to December 2018 concerning 250 selected patients.

DETAILED DESCRIPTION:
As use of inotropes is highly variable between anesthesiologists, the investigators want to study if the choice of the inotropic drugs have an impact on morbid-mortality in paediatric cardiac surgery.

The investigators will retrospectively review the files from patients operated from january 2008 to December 2018. The investigators will concentrate on high risk patients defined as age ≤ 1 year, RACHS score ≥ 3 and complex heart surgery (Switch procedure, atrioventricular canal defect, aortic coarctation or aortic arch interruption, truncus arteriosus, mitral valvuloplasty). The investigators aim for a study population of about 250 patients. Primary outcome will be MODS score defined by death or 2 organ dysfunction (circulatory, respiratory or renal failure).

Statistical analysis:

One propensity score will be performed on two groups: Dobu and Milri. After 15 multiple imputations of the datasets using the mice R package, the CBPS R package will be used to perform the propensity score, estimating an Average Treatment Effect (ATE), using covariate balancing and requesting an exact match, which has been showed to be superior to traditional logistic regression approaches and boosted classification and regression trees . An absolute standardized difference less than 10-15% will be considered to support the assumption of balance between the groups because it is not affected by the sample size, unlike P-values, and it may be used to compare the relative balance of variables measured in different units. The mean and standard deviation obtained after matching for continuous variables, and the percentage for categorical variables will be presented. After the propensity score, the investigators will use the survey R package to perform logistic regressions for binary outcome variables and linear regressions for continuous outcomes, which will include the treatment group effect, the weight resulting from the matching and variables present in the propensity score in order to obtain a doubly-robust estimator which will correct the last remaining possible imbalance between the covariates and produces an unbiased treatment effect. The survey R package includes the Huber-White corrected standard errors, which maintains the standard errors unbiased even under heterogeneity of the residuals. Last, the advantage of a doubly-robust estimator is that it needs only one of the two models (propensity score and logistic regression after the propensity score) to be correctly specified. The so-called 'within approach', that is averaging the treatment effects on the 15 logistic and linear regressions has been showed to produce less biased estimates than the 'Across approach' - that is, performing linear or logistic regressions on averaged imputed matched datasets - especially when missing data is related to the treatment group. The R software (R Core Team, 2019), version 3.6.2. will be used to produce the results.

ELIGIBILITY:
Inclusion Criteria:

Patient under 1 year old. Cardiac surgery with CPB between 2008-2018. RACHS-1 risk categories >3.

We selected the most relevant and common surgery in our center:

* Transposition of the great arteries
* Atrio-ventricular canal defect
* Aortic coarctation or interruption
* Truncus arteriosus
* Mitral valvuloplasty

Exclusion Criteria:

* None

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children under 1 year undergoing complex cardiac surgery with cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
MODS2 score | Weaning from cardiopulmonary bypass in the operating room
  Impact of the inotropic plan on the morbi-mortality. Use of the MODS2 score who is defined by death or 2 organ's failures: circulation, respiratory or renal

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Universitaire des Enfants Reine Fabiola, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No